CLINICAL TRIAL: NCT06667531
Title: Influence of Intermediate Abutment Height and Timing of Placement on Peri-implant Marginal Bone Loss in Single Implant-supported Crowns: a 12-month Follow-up Randomized Clinical Trial.
Brief Title: Evaluation of Marginal Bone Loss (MBL) 12 Months Post-loading of Implants Supporting Individual Crowns, Based on the Height of the Intermediate Abutment and Its Placement Time. Immediate Abutments of 2 or 3 Mm Show the Lowest MBL, Whereas 1.5 Mm or Delayed Abutments Are Associated with Higher MBL.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quintas Hijós Clínica Dental (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Principal Investigator, Jacobo Quintas Hijós, Medical Director, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.I. PI22/324
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Marginal Bone Loss
Keywords: marginal bone loss; abutment height; abutment placement timing
MeSH Terms: interventions — Drug Implants; Surgery, Oral

STUDY DESIGN:
Intervention Model Description: This controlled clinical trial aims to evaluate changes in peri-implant marginal bone levels during the first year of function around platform-switched implants placed 1.5 mm subcrestally and connected to intermediate abutments of heights 1.5, 2, and 3 mm, placed immediately at the time of the first surgery or delayed at the time of the second surgery.
  54 patients received at least one single screw-retained crown on an implant replacing a posterior tooth (60 implants). The implants were divided into six treatment groups based on the height (1.5 mm; 2 mm; 3 mm) and timing of placement (immediate: surgery 1; delayed: surgery 2) of the intermediate abutment: group 1 (height 3; surgery 1), group 2 (height 2; surgery 1), group 3 (height 1.5; surgery 1), group 4 (height 3; surgery 2), group 5 (height 2; surgery 2), group 6 (height 1.5; surgery 2). Mesial and distal linear radiographic measurements (from the implant shoulder to the bone crest) were performed at five follow-up times: implant
Who Masked: Participant, Investigator
Masking Description: Immediately after the placement of the implant, the subject was randomly assigned to one of the six treatment groups by opening a numbered sealed envelope from a computer-generated randomization list. Consequently, the surgeon was unaware of each subject's group assignment until the implant was installed. From that point onward, based on the random assignment, the intermediate abutments of the three heights were screwed with a torque lower than the implant insertion torque to the internal connection either immediately during the same installation procedure (one-abutment-one-time protocol) or delayed during the second surgery procedure at 8 weeks after the installation (two-stage protocol: submerged implant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (height 3; surgery 1) (Active Comparator): Placement of an immediate intermediate abutment (in implant placement surgery). This abutment has a height of 3 mm.
  Interventions: Procedure: Implant
- Group 2 (height 2; surgery 1) (Active Comparator): Placement of an immediate intermediate abutment (in implant placement surgery). This abutment has a height of 2 mm.
  Interventions: Procedure: Implant
- Group 3 (height 1.5; surgery 1) (Active Comparator): Placement of an immediate intermediate abutment (in implant placement surgery). This abutment has a height of 1.5 mm.
  Interventions: Procedure: Implant
- Group 4 (height 3; surgery 2) (Active Comparator): Placement of a delayed intermediate abutment (in the second implant surgery). This abutment has a height of 3 mm.
  Interventions: Procedure: Implant
- Group 5 (height 2; surgery 2) (Active Comparator): Placement of a delayed intermediate abutment (in the second implant surgery). This abutment has a height of 2 mm.
  Interventions: Procedure: Implant
- Group 6 (height 1.5; surgery 2) (Active Comparator): Placement of a delayed intermediate abutment (in the second implant surgery). This abutment has a height of 1.5 mm.
  Interventions: Procedure: Implant

INTERVENTIONS:
Procedure: Implant — Placement of an immediate intermediate abutment (in implant placement surgery). This abutment has a height of 3 mm.
  Other Names: Oral Surgery
  Arms: Group 1 (height 3; surgery 1)
Procedure: Implant — Placement of an immediate intermediate abutment (in implant placement surgery). This abutment has a height of 2 mm.
  Other Names: Oral Surgery
  Arms: Group 2 (height 2; surgery 1)
Procedure: Implant — Placement of an immediate intermediate abutment (in implant placement surgery). This abutment has a height of 1.5 mm.
  Other Names: Oral Surgery
  Arms: Group 3 (height 1.5; surgery 1)
Procedure: Implant — Placement of a delayed intermediate abutment (in the second implant surgery). This abutment has a height of 3 mm.
  Arms: Group 4 (height 3; surgery 2)
Procedure: Implant — Placement of a delayed intermediate abutment (in the second implant surgery). This abutment has a height of 2 mm.
  Arms: Group 5 (height 2; surgery 2)
Procedure: Implant — Placement of a delayed intermediate abutment (in the second implant surgery). This abutment has a height of 1.5 mm.
  Arms: Group 6 (height 1.5; surgery 2)

SUMMARY:
Objectives:To determine which combination of abutment height and timing of placement is most effective in reducing marginal bone loss (MBL).

Materials and Methods: 54 patients received at least one single screw-retained crown on an implant replacing a posterior tooth (60 implants). The implants were divided into six treatment groups based on the height (1.5 mm; 2 mm; 3 mm) and timing of placement (immediate: surgery 1; delayed: surgery 2) of the intermediate abutment: group 1 (height 3; surgery1), group 2 (height 2; surgery1), group 3 (height 1.5; surgery1), group 4 (height 3; surgery2), group 5 (height 2; surgery2), group 6 (height 1.5; surgery2). Mesial and distal linear radiographic measurements (from the implant shoulder to the bone crest) were performed at five follow-up times: implant surgery, crown placement (T1), and at 3 (T2), 6 (T3), and 12 months after loading (T4). Partial and total MBL were compared among the treatment groups.

DETAILED DESCRIPTION:
All installed implants were BTI UnicCa® implants with a flat tetragonal internal connection (BTI Implant System, Vitoria, Spain) of universal (4.1 mm) or wide (5.5 mm) diameter. On all implants, anti-rotational intermediate abutments Ti Golden® UNIT (BTI Implant System, Vitoria, Spain) of universal (4.1 mm) or wide (5.5 mm) width and 1.5 mm, 2.0 mm, or 3.0 mm height were connected, either immediately during the installation surgery (protocol in one phase: one abutment - one time) or delayed during the second surgery procedure 8 weeks after installation (protocol in two phases: submerged implant). (Figure 1). For all patients, standardized digital intraoral radiographs with a silicone key and Rhin ring positioner were recorded during the surgical installation of the implant (baseline), during the placement of the prosthetic crown (8 weeks after surgery), and at 3, 6, and 12 months after prosthetic loading.

* Surgical Procedures. Patients received a complete clinical (periodontal chart) and radiographic (intraoral radiographs, orthopantomography, and CBCT) examination. All surgical procedures were performed by the same surgeon (JQH) under local anesthesia (Artinibsa®; Inibsa Dental SLU, Barcelona, Spain). The implant size was selected based on digital planning with CBCT (Planmeca Romexis Software) according to the quantity and quality of bone. Prior to surgery, the thickness of the soft tissue (from the mucosal surface to the crestal bone) at the implant placement site was measured with a periodontal probe (15 mm, PCP UNC 15; HuFriedy). A conventional placement protocol was followed, with delayed installation of the implant in a fully healed socket (minimum 16 weeks of healing after tooth extraction). Osteotomy was performed without irrigation at low revolutions (100 rpm) following the defined protocol according to implant size and bone density. All implants were placed 1.5 mm subcrestally. All patients received pharmacological prescription with antibiotics (Amoxicillin 1 g every 12 hours for 7 days) or clindamycin in case of allergy, anti-inflammatory medication (Dexketoprofen 25 mg every 8 hours for 3 days), and probiotics (1 sachet per day for 1 week), in addition to postoperative care instructions: pressure with gauze for 5 minutes, application of ice for 10 minutes, soft and cold diet for the first 24 hours, and rinses with 0.12% chlorhexidine (Perioaid; Dentaid SL; Cerdanyola, Spain) twice a day for 7 days. Sutures were removed after 7 days.
* Restorative Procedures. Eight weeks after the implant installation surgery, the platforms of the submerged implants were exposed and the intermediate abutment was connected with a torque of 35 Ncm. Ten weeks after surgery and after increasing the intermediate abutment torque to 35 Ncm on the non-submerged implants, the prosthetic phase began for all cases. All definitive implant-supported prostheses were unitary screw-retained metal-ceramic crowns. Records for the laboratory were obtained in all cases through digital intraoral scanning (iTero®; Align Technology Inc; San José; California, USA). The CAD design of the restorations was done using Exocad Software. The CAM fabrication of the restorations involved milling the metal framework and layering the ceramic covering on a printed model. The unitary crowns were screwed in 2 weeks after the scanning phase with a prosthetic screw torque of 20 Ncm (conventional loading for all cases: 12 weeks after implant placement surgery). The screw channels were sealed with Teflon and compact composite (GrandioSo; Voco GmbH; Cuxhaven, Germany). Occlusion was adjusted, and the adequacy of contact points and gingival sealing was checked.
* Radiographic Evaluation. Standardized digital intraoral radiographs with a silicone key and Rhin ring positioner (Planmeca Prox + Planmeca Prosensor HD; Planmeca Oy; Helsinki, Finland) were obtained at implant placement (baseline), at definitive crown placement (T1), and at 3 months (T2), 6 months (T3), and 12 months (T4) after functional loading. For MBL measurement, the Planmeca Romexis dental imaging software platform was used. Linear measurements were taken in each intraoral radiograph from the most mesial and distal point of the implant shoulder to the crestal bone. The magnification of the radiographs was corrected based on the radiographic measurement of the height and width of each implant, from which each linear MBL measurement was calibrated and recalculated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults.
* Plaque and bleeding indices below 10%.
* Absence of chronic periodontal diseases (periodontitis) or acute periodontal diseases (periodontal abscess).
* Presence of intact alveolar walls.
* Sufficient bone height and width.
* Need for restoration of a tooth in the posterior maxillary or mandibular region (premolars and molars).
* Incorporation into a periodontal maintenance program.

Exclusion Criteria:

* History of systemic disease or radiotherapy contraindicating bone surgery.
* Pregnant or breastfeeding women.
* Smokers of more than 10 cigarettes per day.
* Parafunctional habits.
* Alcohol or drug abuse.
* Narrow interproximal spaces (less than 9 mm).
* Placement of implants flapless or post-extraction.
* Insertion torque during implant placement below 35 Ncm.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss (MBL) measured in mm (mm) 12 months after loading the implant. | 12 months
  Cumulative MBL after 12 months of prosthetic loading measured in millimeters.

SECONDARY OUTCOMES:
Evolution over time of marginal bone loss (MBL) measured in millimeters (mm) at different stages. | 0, 3, 6, 12 months.
  Partial MBL on the day of crown placement and 3, 6 and 12 months after loading, measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Pérez Pevida, Dentistry, Study Director — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

REFERENCES:
- [Derived] Quintas-Hijos J, Perez-Pevida E. Influence of intermediate abutment height and timing of placement on marginal bone loss in single implant-supported crowns: a 12-month follow-up randomized clinical trial. Clin Oral Investig. 2025 May 8;29(6):291. doi: 10.1007/s00784-025-06364-8. PMID 40335732